CLINICAL TRIAL: NCT00586560
Title: A Phase 1 Trial of Escalating Doses of Karenitecin Plus Cyclophosphamide Administered Intravenously Daily for 5 Consecutive Days in Pediatric Patients With Refractory or Recurrent Solid Tumors
Brief Title: Karenitecin in Pediatric Patients With Refractory or Recurrent Solid Tumors N10010)
Acronym: KTN10010
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Pediatric Brain Tumor Consortium (Network)
Responsible Party: Principal Investigator, Susan Blaney, Principal Investigator, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-20159; KTN10010; BMP1350
Record Dates: First submitted 2007-12-20; First posted 2008-01-04 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Solid Tumors
Keywords: solid tumors
MeSH Terms: interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Stratum 1 (~ 25 patients) will include patients with known bone marrow metastases or those who have had prior intensive myelosuppression therapy (including autologous or allogeneic stem cell rescue [SCR], total body irradiation [TBI], craniospinal irradiation [CSI], or hemipelvic radiation).
  Interventions: Drug: Kareniticin and cyclophosphamide
- 2 (Experimental): Stratum 2 (~ 25 patients) will include patients without previous intensive myelosuppressive therapy and bone marrow metastases.
  Interventions: Drug: Kareniticin and cyclophosphamide

INTERVENTIONS:
Drug: Kareniticin and cyclophosphamide — An accelerated titration dose escalation design will be used in this study. Dose escalation will function independently for each stratum. Patients in both strata will receive Karenitecin and cyclophosphamide administered as an IV infusion each day for 5 consecutive days. In addition, patients in Stratum 1 will receive prophylactic G-CSF starting 24 hours after completion of the fifth dose of Karenitecin and cyclophosphamide (and continuing daily until the ANC is over 1500/mm3 after nadir). The regimen will be repeated every 21 days (1 treatment cycle).
  Treatment may continue for up to 20 cycles, provided there is continued evidence of clinical benefit and absence of unacceptable toxicity.

SUMMARY:
This is a Phase 1, open-label, single-center, dose-escalating study in pediatric patients with refractory or recurrent solid tumors. Patients will be registered into 1 of 2 strata, depending upon the presence bone marrow metastases or previous treatment with intensive myelosuppression therapy. Patients will receive Karenitecin along with cyclophosphamide daily for 5 consecutive days, every 21 days (1 treatment cycle). Treatment may continue for up to 20 cycles, as long as there is continued evidence of clinical benefit and an absence of unacceptable toxicity.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, dose-escalating study of karenitecin plus cyclophosphamide in the treatment of pediatric patients with refractory or recurrent solid tumors. All patients must have histologically documented diagnosis of cancer (solid tumors) refractory to conventional therapeutic modalities or for which no curative treatment exists.

Approximately 50 patients will be registered into the study in one of 2 strata.

Stratum 1 will include patients with known bone marrow metastases or those who have had prior intensive myelosuppression therapy. Stratum 2 will include patients without previous intensive myelosuppressive therapy or bone marrow metastases. Each stratum will accrue patients independently.

The primary endpoint in this study is the MTD and determining the recommended Phase 2 dose level for this study. The MTD will be determined for each stratum independently.

There are 3 defined periods in this study:

Period I (Screening and Registration)

Period II (Active Treatment): An accelerated titration dose escalation design will be used in this study. Dose escalation will function independently for each stratum.

Period III (End of Study): Once treatment has been discontinued, patients will undergo end-of-study procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 12 months and less than or equal to 21 years at the time of registration.
2. Histological documentation of cancer (solid tumors) at initial diagnosis. The requirement for histological verification will be waived for patients with intrinsic brainstem gliomas. Patients with non-Hodgkin's lymphomas or Hodgkin's Disease are considered to have non-hematological malignancies.
3. Current disease state must be one which is refractory to curative therapeutic modalities or for which there is no known curative therapy.
4. Karnofsky score greater than or equal to 60 (patients over 10 years of age) and Lansky score greater than or equal to 60 (patients 10 years of age or less). Performance status scales/scores are provided in Appendix E in full protocol attached in Section S.

   Note: Neurological deficits in patients with CNS tumors must have been stable for a minimum of one week before study entry. Patients who are unable to walk because of paralysis, but who are up in a wheelchair will be considered ambulatory for performance score assessment.
5. Fully recovered from any acute toxic effects of all previous chemotherapy, immunotherapy, biological therapy, or radiotherapy before study entry.
6. At least 90 days must have elapsed after autologous or allogeneic stem cell rescue (SCR) and the start of study treatment. There should be no evidence of active graft versus host disease.
7. At least 7 days must have elapsed since the last administration of non-myelosuppressive chemotherapy, immunotherapy or biological therapy and the start of study treatment.
8. At least 21 days must have elapsed since the completion of myelosuppressive chemotherapy and the start of study treatment (at least 42 days must have elapsed if treated with nitrosourea).
9. At least 14 days must have elapsed since the completion of local palliative external beam radiotherapy (XRT - small port) and the start of study treatment. At least 6 months must have elapsed if prior total body irradiation (TBI), craniospinal XRT, or if radiation to 50% or more of pelvis; and at least 42 days must have elapsed if other substantial bone marrow radiation (20% or more of marrow - see Appendix F).
10. Negative serum or urine pregnancy test (female patients of childbearing potential).
11. Agreed to use an effective contraceptive method, including abstinence (male and female patients of reproductive potential).
12. Adequate bone marrow function, defined as: • Peripheral absolute neutrophil count (ANC) 1000/mm3 or greater. • Platelet count 75,000/mm3 or greater (transfusion independent) for Stratum 1. • Platelet count 100,000/mm3 or greater (transfusion independent) for Stratum 2. • Hemoglobin 8.0 g/dL or greater (may receive red blood cell [RBC] transfusions).
13. Adequate renal function; defined as: •Creatinine clearance or radioisotope glomerular filtration rate (GFR) 70 mL/min/m2 or greater.

    OR

    • Serum creatinine based on age as follows: 5 years or less - 0.8 or less mg/dL over 5 years to 10 years old - 1.0 or less mg/dL over 10 years to 15 years old - 1.2 or less mg/dL over 15 years old - 1.5 or less mg/dL
14. Adequate hepatic function; defined as: • Total bilirubin 1.5 mg/dL or less. • ALT 5 or less x upper limit of normal (ULN) for age. • Albumin 2 g/dL or more.
15. Adequate cardiac function; defined as: • No known history of congestive heart failure. • No uncontrolled medically-important cardiac arrhythmias, including ventricular tachycardia/fibrillation, atrial fibrillation, flutter or idioventricular rhythm.
16. Informed consent must be obtained before any study-specific testing is performed or administration of treatment.

Exclusion Criteria:

1. Are pregnant or breastfeeding.
2. Receiving, or have received growth factors that support platelet count, or white cell number or function within 7 days of screening blood work.
3. Patients with CNS tumors who have not been on a stable or decreasing dose of dexamethasone for the past 7 days at the time of screening.
4. Currently receiving treatment with another investigational therapy.
5. Currently receiving treatment with other anti-cancer agents.
6. Have CNS metastases or malignant leptomeningeal involvement that is rapidly progressive, or have poorly controlled seizures (no more than one seizure/month on anti-epileptic therapy).
7. Have an active infection (including viral, fungal, bacterial, rickettsial, mycobacterial, or parasitic).
8. Are judged by the Investigator to be unlikely to be able to fully comply with the study protocol and/or to complete the study or required study procedures.

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2007-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) levels and recommended Phase 2 dose levels of Karenitecin when administered intravenously for 5 consecutive days with a fixed dose of Cytoxan® | evaluation will extend at least 30 days following the last dose or until toxicities have resolved

SECONDARY OUTCOMES:
Secondary objectives include the assessment of toxicity associated with Karenitecin administered in combination with cyclophosphamide; and the assessment of antitumor activity of Karenitecin administered in combination with cyclophosphamide. | evaluation will extend at least 30 days following the last dose or until toxicities have resolved

CONTACTS AND LOCATIONS:
Overall Officials: Susan Blaney, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States